CLINICAL TRIAL: NCT03592524
Title: Effect of Ramadan Fasting on Muslim Recipients After Living Donor Liver Transplantation: Single Center Study
Brief Title: Effect of Ramadan Fasting on Muslim Recipients After Living Donor Liver Transplantation
Status: Completed | Type: Observational
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Iman Fawzy Montasser, Associate professor of tropical medicine , Ain Shams university, Ain Shams University
Other Study IDs: Ramadan fasting and liver
Record Dates: First submitted 2018-06-22; First posted 2018-07-19 (Actual); Last update posted 2018-07-19 (Actual); Status verified 2018-07

CONDITIONS: Liver Transplantation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Fasting Ramadan — Muslims recipients refrain from eating and drinking anything from dawn until sunset(14-15 hours)

SUMMARY:
The study aimed to assess the possibility of Ramadan fasting and to start protocol of adapting immunosupression regiment and scheduled follow up for patients wishing to fast after liver transplantation (LT).

DETAILED DESCRIPTION:
Very limited data in the literature about how to apply Ramadan fasting in the post liver transplant setting. The timing of Ramadan is changeable according to the lunar year and according to time of down and sunset in each country. In Egypt, for example, Ramadan fasting this year started 17th of May and finished 14th June with average fasting hours of 15-16 hours The study aimed to assess the possibility of Ramadan fasting and to start protocol of adapting immunosupression regiment and scheduled follow up for patients wishing to fast after LT.This prospective study included 45 recipients who underwent LT at Ain Shams Center for Organ Transplant (ASCOT), Cairo, Egypt.

ELIGIBILITY:
Inclusion Criteria:

* • Recipients completed their first year after LDLT

  * Normal liver and renal functions at least in the last 3 months before fasting
  * No reported rejection episodes in the last 6 months before the study
  * Recipients wishing to fast Ramadan
  * Informed consent about the study

Exclusion Criteria:

* • First year of LDLT

  * Recipients transplanted for Budd Chiari syndrome
  * Recipients with vascular stents (hepatic artery , portal vein or hepatic vein stents) requiring long life anticoagulation
  * Creatinine clearance <60 ml/min or serum creatinine >1.5 mg/dl at time of initial enrolment in the study.

Ages: 18 Years to 65 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: patients underwent Living donor liver transplantation
Sampling Method: Non-Probability Sample
Enrollment: 45 (Actual)
Dates: Start 2018-05-17 (Actual); Primary Completion 2018-06-14 (Actual); Study Completion 2018-06-21 (Actual)

PRIMARY OUTCOMES:
Effect of fasting on Allograft function among recipients post liver transplantation | 1 month
  Comparison between pre and post fasting state as regards allograft lfunctions , reflected by measuring AST, ALT(liver enzymes) , serum bilirubin , serum albumin +\_ liver biopsy if rejection is suspected
Effect of fasting Ramadan on renal functions among recipients post liver transplantation | 1 month
  Comparison between fasting and post fasting renal functions ( serum creatinine, Blood urea nitrogen ,serum sodium and potassium
Effect of Ramadan fasting on immunosuppressant trough level in liver transplantation recipients | 1 month
  Comparison between fasting and post fasting immunosuppressant drugs trough levels

SECONDARY OUTCOMES:
Effect of Ramadan fasting on blood pressure Among hypertensive recipients on antihypertensive drugs | 1 month
  For hypertension patients regular monitoring of blood pressure by sphingomanometer for any changes in these parameters on daily bases during the months
Effect of fasting Ramadan on blood sugar control among diabetics recipients | 1 month
  Comparison between fasting and post fasting on blood sugar by daily measures of fasting and 2 hours postprandial blood sugar

CONTACTS AND LOCATIONS:
Locations (1):
- Iman Montasser, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided